CLINICAL TRIAL: NCT07371429
Title: Phase 1, Open-Label, Single Arm (Non-comparator) Study to Evaluate the Pharmacokinetics and Safety of a Single Dose of Oral Gepotidacin in Addition to Antibacterial Standard of Care in Pediatric Participants From 2 to Less Than 12 Years of Age With a Suspected or Confirmed Bacterial Infection or Receiving Prophylaxis With Antibiotics
Brief Title: A Study in Pediatric Participants Aged ≥2 to <12 Years With a Suspected or Confirmed Bacterial Infection or Receiving Prophylaxis Antibiotics
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 222778; 2025-522916-17 (EudraCT Number)
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Urinary Tract Infections
Keywords: Gepotidacin; Antibacterial Standard of Care; Antibiotics; Bacterial Infection; Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections; Bacterial Infections | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gepotidacin plus Standard of care (SOC) (Experimental): Single Arm
  Interventions: Drug: Gepotidacin; Drug: SOC

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin will be administered
Drug: SOC — SOC will be administered

SUMMARY:
The study will be conducted to evaluate how a single oral dose of Gepotidacin is processed in the body over time along with safety monitoring in hospitalized pediatric participants who are receiving a standard of care treatment with antibacterials for a confirmed or suspected infection or for its prevention.

ELIGIBILITY:
Inclusion Criteria:

* Participants having ≥2 to <12 years of age at the time of signing the informed consent/assent and have a body weight >=10 kilograms (kg).
* Participants receiving SoC antibacterial therapy for a confirmed/suspected infection or for prophylaxis AND is able to take a single dose of the powder for oral suspension formulation of gepotidacin after a meal.
* Participants either hospitalized or in an overnight clinic. Participant is expected to be in hospital/clinic for at least 24 hours post administration of study intervention.

Participant has an indwelling venous catheter in place as part of the clinical SoC.

* Male or female according to their reproductive organs at birth.
* Pregnancy testing is required as appropriate for the age, sexual activity, and sexual maturity of pediatric participants and as required by local regulations. Investigator should apply clinical judgment.
* A female participant is eligible to participate if she is a WOCBP who is not pregnant as confirmed by a high sensitivity serum or urine pregnancy test at baseline (Day 1) regardless of current or prior contraception use or abstinence, is not breastfeeding, or is not a WOCBP.
* Participant LAR(s) who has the ability to understand, agree to, and sign the informed consent form before initiation of any protocol-related procedures; participant has the ability to give documented assent.
* Participant and participant's LAR are willing and able to comply with study instructions, study visits, and procedures.

Exclusion Criteria:

* Participants having a BMI-for-age that is less than the 5th percentile or greater than the 95th percentile based on the CDC percentiles [CDC NCHS Growth Charts].
* Participants having a clinically significant medical history, including malignancy, significant chromosome abnormality, neurological disorder or history of seizure (excluding simple febrile seizure), chronic immunosuppressive disease, active tuberculosis or acute hepatitis.
* Participants with serious disease/condition that could be imminently life-threatening (e.g. is clinically/hemodynamically unstable, is septicemic, has severe sepsis, organ failure, requiring ITU care or has clinical laboratory tests either nonstable or anticipated to be nonstable) or the participant is unlikely to survive for the duration of the study period.
* The participant has severe renal organ dysfunction or has known anuria, oliguria, or significant impairment of renal function (creatinine clearance <60 mL/min or clinically significant elevated serum creatinine as determined by the investigator).
* The participant has a significant CV history or based on investigator judgment any clinically significant abnormal ECG reading at Screening/baseline (e.g., prolonged QT syndrome).
* The participant has congenital anomalies of the GI tract, heart or liver, including GI tract abnormalities (obstruction, atresia) and Gl tract immaturity.
* The participant has a history of sensitivity to the study intervention, or components thereof, or a history of a drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates study participation.
* The participant is immunocompromised or has altered immune defenses that may predispose the participant to a higher risk of complications (e.g., uncontrolled diabetes in the judgment of the investigator, transplant recipients (with the exception of cornea and autologous BMT), participants with clinically significant persistent granulocytopenia [absolute neutrophil count <1000/μL], and participants receiving immunosuppressive therapy, including corticosteroid therapy [>20 mg/day prednisolone or equivalent for >1 week, 20 mg/day prednisolone or equivalent for >2 weeks, or prednisolone or equivalent ≥10 mg/day for >6 weeks]). Participants with a known CD4 count of <200 cells/mm3 are to not be enrolled.
* The participant has any of the following medical condition that requires medication that may be impacted by inhibition of acetylcholinesterase, such as:

  * Poorly controlled asthma or obstructive pulmonary disease at baseline and, in the opinion of the investigator, not stable on current therapy.
  * Active peptic ulcer disease
  * Juvenile Parkinson disease
  * Juvenile Myasthenia gravis
* The participant has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention (e.g., ileostomy or malabsorption syndrome).
* The participant plans to use any of the prohibited medications or nondrug therapies from the Baseline Visit through Follow-up Visit at 7 ±3 days after the single dose of study intervention.
* The participant has received a prohibited medication within 14 days or 5 half-lives prior to gepotidacin administration, whichever is longer.
* The participant has been previously enrolled in this study or has previously been treated with gepotidacin.
* The participant has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives prior to gepotidacin administration, whichever is longer.
* The participant, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
* If the child is being breastfed:

  * There is suspicion of current alcohol or substance misuse/abuse in breastfeeding mother.
  * The breastfeeding mother is taking any medication or any substances containing any of the medications included in the prohibited medication list with known or unknown lactation excretion.
* The participant has severe hepatic organ dysfunction.
* The participant has an ALT value >2 × ULN.
* The participant has a total bilirubin >1.5xULN; Participants with Gilbert's syndrome can be included with total bilirubin >1.5xULN as long as direct bilirubin is ≤1.5xULN.
* Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* The participant has congenital long QT syndrome or known prolongation of the QTc interval.
* The participant has uncompensated heart failure.
* The participant has severe left ventricular hypertrophy.
* The participant has a family history of QT prolongation or sudden death or history of sudden infant death in a sibling.
* The participant has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or brady arrhythmia within the last 12 months.
* The participant is taking QT-prolonging drugs or drugs known to increase the risk of TdP per the ww.crediblemeds.org. "Known Risk of TdP" category at the time of the Baseline Visit, which cannot be safely discontinued from the Baseline Visit (Day 1) through 7 (+3) days after the single dose of study intervention; or the participant is taking a strong CYP3A4 inhibitor.
* The participant has a mean triplicate QTc >450 msec or a mean triplicate QTc >480 msec for participants with complete bundle branch block.
* The participant has a documented or recent history of uncorrected hypokalemia within the past 3 months.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-08-23 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
AUC from time zero to the time of the last quantifiable concentration (AUC[0-t]) of gepotidacin | Up to 24 hours post dose (Day 1)
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC[0-inf]) of gepotidacin | Up to 24 hours post dose (Day 1)
Maximum observed plasma concentration (Cmax) of gepotidacin | Up to 24 hours post dose (Day 1)
Apparent oral clearance (CL/F) of gepotidacin | Up to 24 hours post dose (Day 1)
Apparent volume of distribution (Vz/F) of gepotidacin | Up to 24 hours post dose (Day 1)
Terminal phase half-life (t1/2) of gepotidacin | Up to 24 hours post dose (Day 1)

SECONDARY OUTCOMES:
Number of participants with Adverse events (AEs), Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs) | Up to 7 days (±3 days)
Change from baseline in vital signs: Temperature | At 2 hours (±15 mins) post dose on Day 1
Change from baseline in vital signs: Blood Pressure | At 2 hours (±15 mins) post dose on Day 1
Change from baseline in vital signs: Pulse Rate | At 2 hours (±15 mins) post dose on Day 1
Change from baseline in Electrocardiogram (ECG) | At 2 hours (±15 mins) post dose on Day 1

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf